CLINICAL TRIAL: NCT02005133
Title: A Prospective, Observational, Multicentre, 2 Year Study Evaluating the Use of Eylea (Aflibercept) for the Treatment of Neovascular (Wet) Age-related Macular Degeneration in UK NHS Opthalmology Clinics
Status: Terminated | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002AGB16
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Wet age-related macular degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VEGF inhibitor naïve
- VEGF inhibitor prior treated

SUMMARY:
To assess the use of aflibercept over a 2 year period in VEGF inhibitor naive and prior treated wet AMD patients managed in 'real wold' clinic settings.

ELIGIBILITY:
Inclusion Criteria:

- Age greater or equal to 50 years Active choroidal neovascularisation secondary to AMD in one or both eyes which in the opinion of the investigator will benefit from treatment with aflibercept Subject willing and able to provide informed consent

Exclusion Criteria:

- Patients must not have had any prior use of either bevacizumab or aflibercept

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects diagnosed with visual impairment due to wet AMD who are undergoing routine assessment in UK opthalmology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Frequency of aflibercept administration | Up to 1 year
  To assess the frequency of clinic visits over a 1 year period in VEGF inhibitor naive wet AMD patients managed in 'real world' clinic settings.

SECONDARY OUTCOMES:
Frequency of clinic visits | Up to 1 year
  To assess how frequently aflibercept is administered over a 2 year period to VEGF inhibitor naive wet AMD patients managed in 'real world' clinic settings and to determine how frequently these subjects are seen in the clinic.
Aflibercept Administration | Up to 2 years
  To assess how frequently aflibercept is administered over 1 year and 2 year periods to prior treated VEGF inhibitor treated wet AMD subjects managed in 'real world' clinic settings and to determine how frequently these subjects are seen in the clinic.
Changes in visual acuity from baseline | Up to 2 years
  To assess how visual acuity changes over 1 year and 2 year periods in both VEGF inhibitor naive and prior treated wet AMD subjects that receive aflibercept.
Change in central retinal thickness from baseline | Up to 2 years
  To assess how central retinal thickness (CRT) changes as determined by optical coherence tomography OCT) over a 1 year and 2 year period in both VEGF inhibitor naive and prior treated wet AMD subjects that receive aflibercept

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharnmaceuticals, Study Director — Novartis
Locations (17):
- United Kingdom (17):
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Bolton
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Southend
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Uxbridge
  - Novartis Investigative Site, York